CLINICAL TRIAL: NCT05695703
Title: Point Prevalence of Side Strain in Fast Bowlers and Effectiveness of Core Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01402 Siraj ul Haq
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Sport Injury; Sports Physical Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Strength Training Group (Experimental): The participants of core strength training group will perform core strength training for 6 weeks (3 days per week).
  Interventions: Other: Core Strength Training Group
- Conventional Training Group (Active Comparator): The participants of conventional training group will perform conventional exercises for 6 weeks (3 days per week).
  Interventions: Other: Conventional Training Group

INTERVENTIONS:
Other: Core Strength Training Group — The participants of experimental group will perform core strength training regime for 6 weeks (3 days per week). Each exercise session will last for a period of 45 mins, the exercises would be performed in 3 sets of 5 repetitions with 5 seconds hold time and 10 seconds rest between each repetition and a minutes rest in between each set.
  Following exercises would be performed :
  Bridge, Crunch, Plank, Side Plank, Mountain Climb.
  Arms: Core Strength Training Group
Other: Conventional Training Group — The participants of conventional group will perform following exercises :
  Running (10 repetitions X 3 sets), Jogging (10 repetitions X 3 sets), Stretching (10 repetitions X 3 sets)
  Rest between Exercises : 10-15 Seconds Rest between Set of Exercises : 30-60 Seconds Cricketers will receive exercises for 8 weeks. There will be 3 sessions per week.
  Arms: Conventional Training Group

SUMMARY:
To find out the prevalence of side strain in fast bowlers and determine the effectiveness of core strength training in treating side strain

DETAILED DESCRIPTION:
A fast bowler needs to have strong core muscles in order to prevent side strain, which can hider the performance. Variation in deliveries , bowling speed and bowling action can be compromised due to side strain injuries specifically in fast bowlers.

A strong and stable core helps to maintain balance and provide strength while performing repetitive movements such as bowling. Core strengthening program should include exercises that are sports specific, conditioning exercises that focus on anterior and posterior musculature of the trunk and hip.

The aim of this study is to find out the prevalence of side strain in fast bowlers and to incorporate strengthening exercises for core muscles to evaluate its effectiveness for side strain.

ELIGIBILITY:
Inclusion Criteria:

* Male fast bowlers
* Age 14 to 40 years

Exclusion Criteria:

* Athletes who have undergone any surgery
* Anyone with history of chest pain due to cardiopulmonary disorders

Ages: 14 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Core Muscle Strength Test | 6 weeks
  The objective of this evaluation is to monitor the development and improvement of an athlete's core strength and endurance over time.
  We will start in the plank exercise position. This is parallel to the ground with your torso straight and rigid, resting your weight on your toes and forearms.
  Start in the modified press up position elbows and feet on the ground, hold this position for 60 seconds, lift your right arm off the ground, hold this position for 15 seconds.
  Return your right arm to the ground and lift the left arm off the ground, hold this position for 15 seconds, return your left arm to the ground and lift the right leg off the ground, hold this position for 15 seconds, return your right leg to the ground and lift the left leg off the ground, hold this position for 15 seconds, lift your left leg and right arm off the ground.
Sahrmann Core Stability Test | 6 weeks
  The Sahrmann core stability test is a 5-level test used to evaluate the ability of the core muscles to stabilize the spine.

SECONDARY OUTCOMES:
Ultrasonographical assessment of side strain | 6 weeks
  The integration of ultrasound imaging with musculoskeletal modelling has the potential to create new opportunities in the study of human movement science.
  Ultrasound will be performed by scanning in a location immediately inferior to the tender rib in the longitudinal and transverse directions for iden-tification of a muscle tear. The fibers of the internal oblique muscle lie deep in relation to the external oblique muscle fibres and run in a direction different from the external oblique muscle fibres by passing in a superior and medial direction. The internal oblique muscle appears as a sheet of linear fibril-lar echotexture. Tears were defined as loss of the normal fibrillar echotexture pattern with a hypoechoic gap at the rib or costal cartilage attachment of the internal oblique muscle.
Cornell Musculoskeletal Discomfort Questionnaire | 6 weeks
  The Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) was used to assess discomfort. Professor Alan Hedge and Ergonomics students at the Cornell University developed a well-designed data collection tool named CMDQ. The CMDQ is a 54-item questionnaire that includes a body chart and questions about musculoskeletal ache, pain, or discomfort occurrence in 20 parts of the body over the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Saad Rauf, Ph.D*, Principal Investigator — Riphah University
Locations (1):
- Sawar Muhammad Hussain Shaheed Sports Stadium, Gujar Khan, Gujar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No